CLINICAL TRIAL: NCT02490098
Title: An Open-label, Randomized, Five-way, Cross-over Study to Compare the Efficacy of Single- and Dual-hormone Closed-loop Operations Combined With Either Conventional Carbohydrate Counting or a Simplified Qualitative Meal-size Estimation, and Sensor-augmented Pump Therapy in Regulating Glucose Levels in Children and Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Postprandial Glucose Levels in Children and Adults With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-13
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Closed-loop system; Artificial pancreas; Insulin; Glucagon; Hypoglycemia; Postprandial glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Hypoglycemia | interventions — Methods; Insulin; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single-hormone closed-loop strategy with full boluses (Active Comparator): Variable subcutaneous insulin infusion rates will be used to regulate postprandial glucose levels. Patient's usual fast acting insulin analog (Lispro, Aspart or Glulisine) will be infused using a subcutaneous infusion pump (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to the Smartphone platform, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pump. Each subject insulin-to-carbohydrate ratio will be used to calculate the insulin bolus to be given.
  Interventions: Other: 6-day intervention with single-hormone closed-loop strategy; Drug: Insulin; Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic; Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic
- Dual-hormone closed-loop strategy with full boluses (Active Comparator): Variable subcutaneous insulin and glucagon infusion rates will be used to regulate postprandial glucose levels. Patient's usual fast acting insulin analog (Lispro, Aspart or Glulisine) and Glucagon (Eli Lilly) will be infused using two separate subcutaneous infusion pumps (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to the Smartphone platform, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pumps. Each subject insulin-to-carbohydrate ratio will be used to calculate the insulin bolus to be given.
  Interventions: Other: 6-day intervention with dual-hormone closed-loop strategy; Drug: Insulin; Drug: Glucagon; Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic; Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic
- Single-hormone closed-loop strategy with partial boluses (Active Comparator): Variable subcutaneous insulin infusion rates will be used to regulate postprandial glucose levels. Patient's usual fast acting insulin analog (Lispro, Aspart or Glulisine) will be infused using a subcutaneous infusion pump (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to the Smartphone platform, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pump. The partial bolus will be based on the estimated meal size (snack-regular-large-very large). For this strategy, meal size will be defined as: snack as any meal less than 30g, regular meal as any meal between 30g and 60g CHO, large meal as any meal between 60g and 90g CHO, very large meal for anything above 90g CHO. The meal size assessment will be done by the patient.
  Interventions: Other: 6-day intervention with single-hormone closed-loop strategy; Drug: Insulin; Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic; Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic
- Dual-hormone closed-loop strategy with partial boluses (Active Comparator): Variable subcutaneous insulin and glucagon infusion rates will be used to regulate postprandial glucose levels. Patient's usual fast acting insulin analog (Lispro, Aspart or Guilisine) and Glucagon (Eli Lilly) will be infused using two separate subcutaneous infusion pumps (MiniMed® Paradigm® Veo™, Medtronic). Every 10 minutes, the glucose levels as measured by the sensor (Enlite sensor®, Medtronic) will be transferred automatically to the Smartphone platform, that harbors the algorithm, that will calculate the recommended doses and will send it wirelessly to the infusion pumps. The partial bolus will be based on the estimated meal size (snack-regular-large-very large). For this strategy, meal size will be defined as: snack as any meal less than 30g, regular meal as any meal between 30g and 60g CHO, large meal as any meal between 60g and 90g CHO, very large meal for anything above 90g CHO. The meal size assessment will be done by the patient.
  Interventions: Other: 6-day intervention with dual-hormone closed-loop strategy; Drug: Insulin; Drug: Glucagon; Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic; Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic
- Sensor-augmented pump therapy (Active Comparator): Subjects will use sensor-augmented pump therapy and freely implement their usual basal rate and CHO-matching full prandial bolus to regulate glucose levels. Patient's usual fast acting insulin analog will be infused using a subcutaneous insulin infusion pump. Each subject insulin-to-carbohydrate ratio will be used to calculate the insulin bolus to be given.
  Interventions: Other: 6-day intervention with sensor-augmented pump therapy; Drug: Insulin; Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic; Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic

INTERVENTIONS:
Other: 6-day intervention with sensor-augmented pump therapy — One day prior to the intervention, participants will have to install a glucose sensor and the study insulin pump. Participants will adjust their insulin delivery as per their standard practice; including temporary basal and correction boluses. Participants will have access to their finger-stick glucose measurements and will be advised to measure their glucose level as per their standard practice. Participants will be asked to install a new infusion set every 2 days. Participants will be allowed to eat whatever they want and allowed to drink alcohol. Participants will use sensor-augmented pump therapy for 6 days.
  Arms: Sensor-augmented pump therapy
Other: 6-day intervention with single-hormone closed-loop strategy — One day prior to the intervention, participants will have to install a glucose sensor and the study insulin pump. On the first day of the intervention, participants will be admitted to the clinical research facility in the morning. A team member will review with the participant how to use study devices. Competency on the use of study devices will be assessed by a team member. Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be allowed to go home in the afternoon. They will be advised to continue with study intervention at home for the next 5 days. Participants will be asked to install a new infusion set every 2 days. Participants will be allowed to eat whatever they want and allowed to drink alcohol.
  Arms: Single-hormone closed-loop strategy with full boluses; Single-hormone closed-loop strategy with partial boluses
Other: 6-day intervention with dual-hormone closed-loop strategy — One day prior to the intervention, participants will have to install a glucose sensor and the study insulin pump. On the first day of the intervention, participants will be admitted to the clinical research facility in the morning. Participants will have to install a second pump containing glucagon. A team member will review with the participant how to use study devices. Competency on the use of study devices will be assessed by a team member. Only participants demonstrating competency on use of study devices will be allowed to continue to the home study phase. Participants will be allowed to go home in the afternoon. They will be advised to continue with study intervention at home for the next 5 days. Participants will be asked to install a new infusion set every 2 days. Participants will be allowed to eat whatever they want and allowed to drink alcohol.
  Arms: Dual-hormone closed-loop strategy with full boluses; Dual-hormone closed-loop strategy with partial boluses
Drug: Insulin — Participant's usual fast-acting insulin analog will be used: Lispro (Humalog), Aspart (NovoRapid) or Glulisine (Apidra)
Drug: Glucagon — Glucagon (Eli Lilly) will be used during dual-hormone closed-loop strategy.
  Arms: Dual-hormone closed-loop strategy with full boluses; Dual-hormone closed-loop strategy with partial boluses
Device: Continuous Glucose Monitoring System Enlite sensor®, Medtronic — Enlite sensor®, Medtronic
Device: Insulin pump MiniMed® Paradigm® Veo™, Medtronic — MiniMed® Paradigm® Veo™, Medtronic

SUMMARY:
Current intensive insulin therapy in T1D involves prandial insulin boluses depending on the carbohydrate content of each ingested meal. Carbohydrate content of ingested meals is the main determinant of post-meal glucose excursion. Therefore, accurate carbohydrate counting is a critical aspect of managing postprandial blood glucose levels in type 1 diabetes in order to avoid too much or too little insulin resulting in hypoglycemia and hyperglycemia, respectively. Precision of carbohydrate counting is associated with better glycemic control. However, accurate carbohydrate counting is a challenging task for many patients with type 1 diabetes. Recent developments of continuous glucose sensors and insulin infusion pumps have motivated the research toward "closed-loop'' strategies to regulate glucose levels in patients with type 1 diabetes. In a closed-loop strategy, the pump insulin infusion rate is altered based on a computer generated recommendation that rely on continuous glucose sensor readings. A dual-hormone closed-loop strategy has also been recently proposed to regulate glucose levels. In a dual-hormone strategy, subcutaneous insulin delivery is accompanied by subcutaneous glucagon infusion. Postprandial meal glucose control with closed-loop strategy still needs some improvements. The objective of this study is to test in outpatient unrestricted settings whether, in the context of closed-loop strategy, conventional meal carbohydrate counting could be reduced to a simplified qualitative meal size estimation without a significant degradation in overall glycemic control in children and adult patients with type 1 diabetes. The investigators hypothesize that 1) dual-hormone closed-loop strategy with qualitative meal size estimation is equivalent to dual-hormone closed-loop strategy with CHO counting in terms of mean glucose; 2) single-hormone closed-loop strategy with qualitative meal size estimation is equivalent to single-hormone closed-loop strategy with CHO counting in terms of mean glucose;

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 8 years old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months and currently using a fast actin insulin analog (Lispro, Aspart or Guilisine).
4. Last (less than 3 months) HbA1c ≤ 10%.
5. Currently using carbohydrate counting as the meal insulin dose strategy.
6. Live in the area of Montreal

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Pregnancy.
4. Severe hypoglycemic episode within 1 month of screening.
5. Agents affecting gastric emptying (Motilium®, Prandase®, Victoza®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, SGLT-2 inhibitors and DPP-4 inhibitors) if not at a stable dose for 3 months. Otherwise, these medications are acceptable and will be kept stable during the entire protocol.
6. Oral steroids unless patients present a low stable dose (e.g. 10 mg or less of prednisone per day or physiological doses, less than 35 mg/day, of hydrocortisone Cortef®). Inhale steroids at stable dose in the last month are acceptable.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator (e.g. unstable psychiatric condition).
8. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, follow algorithm's suggestions, etc).
9. Living or planned travel outside Montreal (> 1h of driving) area during closed-loop procedures.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Mean day-and-night glucose levels | 6 days

SECONDARY OUTCOMES:
Percentage of time of glucose levels between 4.0 and 8.0 mmol/L | 6 days
Percentage of time of glucose levels between 4.0 and 10.0 mmol/L | 6 days
Percentage of time of glucose levels above 10.0 mmol/L | 6 days
Percentage of time of glucose levels above 14.0 mmol/L | 6 days
Percentage of time of glucose levels spent below 4.0 mmol/L | 6 days
Percentage of time of glucose levels spent below 3.1 mmol/L | 6 days
Area under the curve of glucose values below 4.0 mmol/L | 6 days
Area under the curve of glucose values below 3.1 mmol/L | 6 days
Number of patients with at least one hypoglycemic event below 3.1 mmol/L with or without symptoms | 6 days
Total number of hypoglycemic event below 3.1 mmol/L | 6 days
Total insulin delivery | 6 days
Total glucagon delivery | 6 days
Standard deviation of glucose levels | 6 days
Total carbohydrate intake | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada